CLINICAL TRIAL: NCT07035470
Title: Biological Age as a Prognostic Marker in Hospitalized Patients With Advanced Cancer: A Retrospective Analysis Based on PhenoAge Model
Brief Title: Biological Age Predicts 90-Day Mortality in Advanced Cancer
Acronym: BIOAGE-CAN
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Galip Can Uyar, MD, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK-2025-0149
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumors Cancer; Hospitalizations
Keywords: Biological Age; PhenoAge; Advanced Cancer; Hospitalized Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized Advanced Cancer Patients: Patients hospitalized with advanced solid tumors (Stage III or IV) in the oncology clinic were retrospectively analyzed. Biological age was calculated using the PhenoAge model. Clinical outcomes such as mortality, ECOG score, mCCI, and length of stay were assessed.
  Interventions: Other: PhenoAge-Based Biological Age Assessment

INTERVENTIONS:
Other: PhenoAge-Based Biological Age Assessment — Biological age was retrospectively calculated using the PhenoAge algorithm, based on nine routine laboratory parameters and chronological age. This model estimates phenotypic aging and was used to predict short-term outcomes including mortality, functional status, comorbidity burden, and hospital length of stay. No new intervention was administered; all data were collected from existing medical records.

SUMMARY:
This retrospective study evaluates whether biological age, calculated using the PhenoAge model, predicts short-term outcomes in patients with advanced cancer who were hospitalized. The main goal is to investigate associations between biological age and short-term mortality, functional status (ECOG), comorbidity burden (mCCI), and length of hospital stay. All data were collected from medical records without any patient intervention.

DETAILED DESCRIPTION:
This is a retrospective observational study including hospitalized adult patients with stage III or IV solid tumors admitted to Etlik City Hospital between November 5, 2022 and December 31, 2024. Patients were included if they stayed for ≥48 hours and had all required laboratory values for calculating biological age using the Levine PhenoAge model. The study aimed to evaluate the association between biological age and (1) 30- and 90-day mortality, (2) ECOG performance score, (3) modified Charlson Comorbidity Index (mCCI), and (4) hospital length of stay. Regression and survival analyses were used to identify prognostic factors. All data were anonymized and collected retrospectively from hospital records.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in the Medical Oncology Department between November 5, 2022, and December 31, 2024

Histologically confirmed advanced-stage (stage III-IV) solid tumors

Age ≥18 years

Hospital stay of at least 48 hours

Actively receiving chemotherapy or received it within the last 6 months

Availability of all 9 required laboratory tests (albumin, creatinine, glucose, CRP, lymphocyte %, MCV, RDW, ALP, WBC) for PhenoAge calculation during the first admission

Patients with multiple hospitalizations who meet the inclusion criteria will be included

Exclusion Criteria:

* Elective hospitalizations (e.g., planned chemotherapy, biopsy)

Patients who died during the first admission

Missing required laboratory parameters

ICU patients and unconscious patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study includes adult patients (≥18 years old) with advanced-stage solid tumors who were hospitalized at Etlik City Hospital, Turkey, between November 5, 2022, and December 31, 2024. Only patients with at least 48 hours of hospitalization and complete laboratory data necessary for PhenoAge calculation were included. The study population represents a real-world sample of hospitalized cancer patients at elevated risk of short-term adverse outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 1615 (Actual)
Dates: Start 2022-11-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
90-Day All-Cause Mortality | Up to 90 days post-admission
  All-cause mortality within 90 days following the date of hospital admission (index hospitalization).

SECONDARY OUTCOMES:
Modified Charlson Comorbidity Index (mCCI) | Baseline (Day of hospital admission)
  The Modified Charlson Comorbidity Index (mCCI) is a validated scoring system used to quantify comorbidity burden. It includes 19 comorbid conditions with weighted values and incorporates age adjustment. Scores range from 0 to 33. In this study, age points are added only for patients aged 50 years and above: +1 point for ages 50-59, +2 for 60-69, +3 for 70-79, and +4 for ≥80.
  Higher mCCI scores indicate greater comorbidity burden and are associated with poorer clinical outcomes. The score is calculated retrospectively from documented diagnoses in the medical records at baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No